CLINICAL TRIAL: NCT04330586
Title: A Trial of Ciclesonide to Assess The Antiviral Effect for Adults With Mild-to-moderate COVID-19
Brief Title: A Trial of Ciclesonide in Adults With Mild-to-moderate COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Woo Joo Kim, Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KUMC-COVID-19
Record Dates: First submitted 2020-03-31; First posted 2020-04-01 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Ciclesonide; Viral load; Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — ciclesonide

STUDY DESIGN:
Intervention Model Description: This multicenter study is an open-labelled, randomized clinical trial for 1:1 ratio of ciclesonide or control arm (standard care)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ciclesonide (Experimental): Ciclesonide 320ug oral inhalation q12h for 14 days
  Interventions: Drug: Ciclesonide Metered Dose Inhaler [Alvesco]
- Control (No Intervention): Standard care without ciclesonide

INTERVENTIONS:
Drug: Ciclesonide Metered Dose Inhaler [Alvesco] — Ciclesonide 320ug oral inhalation q12h for 14 days
  Arms: Ciclesonide

SUMMARY:
According to In vitro studies, ciclesonide showed good antiviral activity against severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). Although some cases were reported for the clinical effectiveness of ciclesonide in the treatment of COVID-19, there is no clinical trial to evaluate the antiviral effect on the reduction of viral load in patients with COVID-19. In this study, we aimed to investigate whether ciclesonide inhalation could eradicate SARS-CoV-2 compared to standard supportive care in patients with mild COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild COVID-19 (NEWS scoring system 0-4)
* Patient within 7 days from symptom onset or Patient within 48 hous after laboratory diagnosis (SARS-CoV-2 RT-PCR)

Exclusion Criteria:

* Hypoxia (SaO2 <95%)
* Unable to take oral medication
* Unable to use inhaler
* Pregnancy or breast feeding
* Immunocompromising conditions
* Moderate/severe renal dysfunction : creatinine clearance (CCL) < 30 mL/min
* Moderate/severe liver dysfunction: AST or ALT > 5 times upper normal limit
* Asthma or chronic obstructive lung disease

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Rate of SARS-CoV-2 eradication at day 14 from study enrollment | Hospital day 14
  Viral load

SECONDARY OUTCOMES:
Rate of SARS-CoV-2 eradication at day 7 from study enrollment | Hospital day 7
  Viral load
Time to SARS-CoV-2 eradication (days) | Hospital day 1, 4, 7, 10, 14, 21
  Viral load
Viral load area-under-the-curve (AUC) reduction versus control | Hospital day 1, 4, 7, 10, 14, 21
  Viral load change
Time to clinical improvement (days) | Up to 28 days
  Resolution of all systemic and respiratory symptoms for ≥2 consecutive days
Proportion of clinical failure | Up to 28 days
  High-flow oxygen therapy or mechanical ventilation requiring salvage therapy

OTHER OUTCOMES:
Safety and tolerability of study drug | Up to 28 days
  Number of adverse events, proportion of early discontinuance

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Song JY, Yoon JG, Seo YB, Lee J, Eom JS, Lee JS, Choi WS, Lee EY, Choi YA, Hyun HJ, Seong H, Noh JY, Cheong HJ, Kim WJ. Ciclesonide Inhaler Treatment for Mild-to-Moderate COVID-19: A Randomized, Open-Label, Phase 2 Trial. J Clin Med. 2021 Aug 12;10(16):3545. doi: 10.3390/jcm10163545. PMID 34441840
- [Derived] Farne H, Singanayagam A. Reply. J Allergy Clin Immunol. 2021 Mar;147(3):1117-1118. doi: 10.1016/j.jaci.2020.11.019. Epub 2020 Dec 30. No abstract available. PMID 33388170
- [Derived] Nicolau DV, Bafadhel M. Inhaled corticosteroids in virus pandemics: a treatment for COVID-19? Lancet Respir Med. 2020 Sep;8(9):846-847. doi: 10.1016/S2213-2600(20)30314-3. Epub 2020 Jul 30. No abstract available. PMID 32738928